CLINICAL TRIAL: NCT07068386
Title: Implementation of Telerehabilitation Includes Neuromotor Assessment and Early Intervention for Preterm Infants
Brief Title: Telerehabilitation for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aysu Kahraman, Assistant Professor (Ph.D.), Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021/219
Record Dates: First submitted 2025-05-28; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Early Intervention; Infant, Premature; Telerehabilitation
Keywords: Early intervention; infant; premature; telerehabilitation
MeSH Terms: conditions — Premature Birth | interventions — Early Intervention, Educational; Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infant (Experimental): The study was conducted using a single-arm design to investigate the feasibility and short-term effectiveness of early intervention delivered via telerehabilitation on the gross motor development of preterm infants. The intervention was individualized for each infant, based on principles of typical motor development, motor learning, and environmental enrichment
  Interventions: Other: Early intervention with telerehabilitation

INTERVENTIONS:
Other: Early intervention with telerehabilitation — All premature infants aged 3 to 5 months included in the study were assessed for motor development using the General Movements Assessment (GMs) and the Alberta Infant Motor Scale (AIMS), based on videos submitted by their parents. Following the video evaluations, parents were contacted via video call. An intervention program was developed in collaboration with the parents, guided by the video-based assessments.
  The intervention program focused on the acquisition of age-appropriate motor development and included components such as massage, positioning, trunk control, movement selectivity, and anti-gravity activities. It was delivered to parents through synchronous. Parents were advised to implement the program for 30 minutes per day, 4 days a week, over a 12-week period. After the intervention, the infants were re-evaluated using the AIMS via video call.

SUMMARY:
The aim of this study is to investigate the feasibility and short-term effectiveness of early intervention delivered via telerehabilitation on the gross motor development of preterm infants.

The motor development of preterm infants will be assessed through video recordings. Based on these assessments and in collaboration with the parents, an intervention program will be developed. The parents will implement this intervention with their infants over a three-month period. Following this, motor development will be reassessed via video recordings.

ELIGIBILITY:
Inclusion Criteria:

* Between November 2021 and May 2024, all preterm infants with a corrected age of 3 to 5 months who were referred to the our Department were invited to participate in the study.

Exclusion Criteria:

* Infants with genetic abnormalities, hospitalized infants, those with blindness or deafness, infants requiring respiratory support, and physiologically unstable infants were excluded from the study.
* Additionally, infants whose parents did not have the required technological equipment for telerehabilitation (mobile phone) or the skills to use it were not included in the study.
* Children with optimal MOS-R were excluded from the study

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Motor Optimality Score-Revised (MOS-R) - A numerical result is obtained by observing the spontaneous motor movements, movement pattern, age adequate movement repertoire, postural patterns and movement character of infants. | MOS-R will be administered on Day 1 (baseline). If the baseline MOS-R score is ≤14, the MOS-R will be repeated on Days 8, 15, 22, and 29. If the score is greater than 14, no further MOS-R assessments will be performed.
  The infant's spontaneous motor movements in the fidgety period (corrected 3-5 months) are recorded on video for 3-5 minutes. The infant must be active and awake, and no external stimuli should be provided. The MOS-R is made with Gestalt perception on this recording.
  MOS-R consists of the sum of five subcategories. Spontaneous motor movements (normal=12, abnormal=4, absent=1 point), movement pattern (normal>abnormal=4, normal=abnormal=2 point, normal<abnormal=1 point), age adequate movement repertoire (present=4, reduced=2, absent=1 point), postural patterns (normal>abnormal=4, normal=abnormal=2, normal<abnormal= 1 point) and movement character (smooth and fluent=4, abnormal=2, cramped synchronized=1 point) The MOS-R ranges from 5 to 28, with higher scores indicating better outcomes. A score between 25 and 28 is considered optimal, 20 to 24 is mildly reduced, 9 to 19 is moderately reduced, and 5 to 8 is severely reduced.
Alberta Infant Motor Scale (AIMS) - A numerical value is obtained by observing the child's gross motor development in the prone, supine, sitting and standing positions. | AIMS will be administered twice: once at baseline (Day 1) and once 13 weeks after baseline.
  It is a norm-referenced tool that evaluates the gross motor development of infants between 0-18 months. This tool evaluates weight transfer, posture and movement against gravity in prone, supine, sitting and standing positions.
  The infant receives a score between 0 and 58, depending on age. This score is then converted to a percentile. A higher percentile mean a better outcome.

OTHER OUTCOMES:
Characteristics of infants and mothers | It will be recorded at study baseline.
  Gestational age (week)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Birth weight (gram)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Gender (female/male)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Multiple pregnancy (single/twin)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Maternal age (year)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Maternal education (primary/high/higher school)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Number of siblings (number)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Duration of hospital (day)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Respiratuar distress syndrome (yes/no)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Preeclampsia (yes/no)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Seizure (yes/no)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Intracranial hemorrhage (yes/no)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Retinopathy of prematurity (yes/no)
Characteristics of infants and mothers | It will be recorded at study baseline.
  Economic status (low/moderate/high)

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the results will be analyzed from the infants' whole body images, it will not be appropriate to share the data.

REFERENCES:
- [Background] Schlichting T, Martins da Silva K, Silva Moreira R, Marques de Moraes MV, Cicuto Ferreira Rocha NA, Boyd RN, Neves Dos Santos A. Telehealth Program for Infants at Risk of Cerebral Palsy during the Covid-19 Pandemic: A Pre-post Feasibility Experimental Study. Phys Occup Ther Pediatr. 2022;42(5):490-509. doi: 10.1080/01942638.2022.2057209. Epub 2022 Mar 27. PMID 35341469